CLINICAL TRIAL: NCT05075031
Title: Could Docosahexaenoic Acid (DHA), Contained in Breast Milk and Artificial Baby Milks, Protect Infants and Children From COVID-19 and Make Them Less Prone to COVID-19-related Severe Illness Than Adults?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kafrelsheikh University (Other)
Collaborators: Ministry of Health, Saudia Arabia (Unknown)
Responsible Party: Principal Investigator, Mahmoud Ramadan mohamed Elkazzaz, Clinical Scientist, Kafrelsheikh University
Other Study IDs: Observational COVID-19 Study
Record Dates: First submitted 2021-10-06; First posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: COVID19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 300 Newborn feeding on Breast Milk or Artificial Milk Formula rom birth to about 2 months of age: The electronic patient record of 300 Newborn feeding on Breast Milk or Artificial Milk Formula from birth to about 2 months of age would be examined and followed between March 2020 and October 2021 and compare their rates of Covid-19 infection, hospitalization and complications with the rates of the Control Groups
- 300 Infant feeding on Breast Milk or Artificial Milk Formula from 2 months to 1 year: The electronic patient record of 300 Infant feeding on Breast Milk or Artificial Milk Formula from 2 months to 1 year would be examined and followed between March 2020 and October 2021 and compare their rates of Covid-19 infection, hospitalization and complications with the rates of the rates of the Control Groups
- 300 child feeding on Breast Milk or Artificial Milk Formula from 1 year to 5 year: The electronic patient record of 300 child feeding on Breast Milk or Artificial Milk Formula from 1 year to 5 year would be examined and followed between March 2020 and October 2021 and compare their rates of Covid-19 infection, hospitalization and complications with the rates of the rates of the Control Groups
- 300 child feeding on Breast Milk or Artificial Milk Formula from 5 year up to 15 year: The electronic patient record of 300 child feeding on Artificial Milk Formula or any source of DHA from 5 year up to 15 year would be examined and followed between March 2020 and October 2021 and compare their rates of Covid-19 infection, hospitalization and complications with the rates of the Control Groups
- Control Group: 1. The electronic patient record of 150 infant and child patients who feed on only cow's milk which does not provide a rich source of DHA and did not feed on any Artificial Milk Formula or any source of DHA would be examined and followed between March 2020 and October 2021 and compare their rates of Covid-19 infection, hospitalization and complications with the rates of the cohorts that feed on Breast Milk or Artificial Milk Formula
  2. The electronic patient record of 150 adult patients from 15 years to 25 years who did not feed on any Artificial Milk Formula or any source of DHA would be examined and followed between March 2020 and October 2021

SUMMARY:
Could Docosahexaenoic Acid (DHA) Protect Infants and Children From COVID-19 and Make Them Less Susceptible to COVID-19-related Severe Illness Than Adults?

* The study is configured as a retrospective and prospective observational study. The study will be multi-center and will involve all Infants and Children feeding on breast milk or Artificial milk formula that contained on DHA.
* Human milk is the best form of infant nutrition providing significant protection against many illnesses for term and preterm infants.
* This study seeks to investigate the possible protective role of DHA found in Breast Milk or Artificial Milk Formula that are used for feeding of Children and Infants.
* This study would examine the electronic patient record of Newborn from birth to about 2 months of age and Infants from 2 months to 1 year old as well as children from 1year to age 5 years old , feeding on Breast Milk or Artificial Milk Formula between March 2020 and October 2021 and compare their rates of Covid-19 infection, hospitalization and complications with the rates of the local age-matched background population.
* As Covid-19 is a new disease, the existing research literature on this specific topic is extremely limited, and so far this study would be the first in this area.

Abstract

The novel SARS-CoV-2, which causes the disease called COVID-19, has rapidly spread across the globe. A striking and consistent observation has been the difference in severity of COVID-19 at different ages: severity, the need for hospitalization and mortality rise steeply with older age while severe disease and death are relatively rare in children and young adults. Most children infected with SARS-CoV-2 are asymptomatic or have mild symptoms, most commonly fever, cough, pharyngitis, gastrointestinal symptoms and changes in sense of smell or taste. Whether children are also less often infected by SARS-CoV-2 is an ongoing debate. Large epidemiological studies suggest that children comprise only 1 to 2% of all SARS-CoV-2 cases. However, these numbers heavily depend on testing criteria and, in many reports, testing was done only in individuals who were symptomatic or required hospitalisation, which is less often the case for children. Some studies suggest that children are just as likely as adults to become infected with SARS-CoV-2.9 However, more recent studies report that children are less likely to get infected after contact with a SARS-CoV-2-positive individual.10-14 It has been suggested that children and adolescents have similar viral loads and may therefore be as likely to transmit SARS-CoV-2 as adults. In addition, the viral load may be similar in asymptomatic and symptomatic individuals. However, reassuringly, transmission in schools from children either to other children or to adults has been rare. The observation that children are less often infected with SARS-CoV-2 and that they have less severe symptoms is similar to that reported for SARS-CoV-1 and Middle East respiratory syndrome (MERS)-CoV. However, this pattern is strikingly different to that for infection with most other respiratory viruses (eg, respiratory syncytial virus (RSV), metapneumovirus, parainfluenza or influenza viruses), for which the prevalence and severity are both higher in children. Dr Amr kamel khalil Ahmed and Dr. Mahmoud Elkazzaz, the lead investigators of this observational study , recently published a preprint that demonstrated Docosahexaenoic acid (DHA) had a high binding affinity and greatest interactions with ACE2 active sites, as well as a moderate binding affinity and moderate interactions with the active sites of IL-6. The Docosahexaenoic acid (DHA) interacts with different active sites of IL6 and ACE2 which are involved in direct or indirect contacts with the ACE2 and IL-6 receptors which might act as potential blockers of functional ACE2 and IL-6 receptor complex. Docosahexaenoic acid (DHA) was detected in abundance in breast milk and other algal sources milk supplement used for newborns and children's feeding. As a result, we believe that docosahexaenoic acid (DHA) may protect children and newborns thorough competing with COVID-19 for ACE2 receptors and inhibiting IL-6 activity and may possibly help them avoid a cytokine storm and save their lives through inhibiting IL-6 and preventing SARS-CoV-2 RBD attachment to ACE2

DETAILED DESCRIPTION:
The study is configured as a retrospective and prospective observational study. The study will be multi-center and will involve all Infants and Children feeding on breast milk or Artificial milk formula that contained on DHA.

Human milk is the best form of infant nutrition providing significant protection against many illnesses for term and preterm infants.

Docosahexaenoic acid (DHA) was detected in abundance in breast milk and other algal sources milk supplement used for newborns and children's feeding. DHA concentration in breast milk varies more than 20-fold across human populations (0.06-1.4% by weight).

Naturally, cow's milk does not provide a rich source of DHA however in most companies whole milk and partially skimmed milk (2%) are fortified with DHA by adding DHA rich feed additive to Market milk formula. Therefore, we will take a cohort of children and infants who feed on natural cow's milk without any processing not breast milk or Artificial milk formula contained on DHA additive as a control.

More recent studies report that children are less likely to get infected after contact with a SARS-CoV-2-positive individual.10-14 It has been suggested that children and adolescents have similar viral loads and may therefore be as likely to transmit SARS-CoV-2 as adults. Therefore, we will take a cohort of adults who did not feed on any Artificial milk formula contained on DHA additive as a control.

This study seeks to investigate the possible protective role of DHA found in Breast Milk or Artificial Milk Formula that are used for feeding of Children and Infants.

This study would examine the electronic patient record of Newborn from birth to about 2 months of age and Infants from 2 months to 1 year old as well as children from 1year to age 5 years old , feeding on Breast Milk or Artificial Milk Formula between March 2020 and October 2021 and compare their rates of Covid-19 infection, hospitalization and complications with the rates of the local age-matched background population.

As Covid-19 is a new disease, the existing research literature on this specific topic is extremely limited, and so far this study would be the first in this area.

ELIGIBILITY:
Inclusion Criteria:

1. Newborn feeding on Breast Milk or Artificial Milk Formula from birth to about 2 months of age.
2. Infant feeding on Breast Milk or Artificial Milk Formula from 2 months to 1 year
3. Children feeding on Breast Milk or Artificial Milk Formula from 1 year to 5 year.
4. Children feeding on Breast Milk or Artificial Milk Formula from 5 year up to 15 year
5. Adult patients from 15 years to 25 years who did not feed on any Artificial Milk Formula or any source of DHA .
6. Infants and children patients who feed on only cow's milk which does not provide a rich source of DHA and did not feed on any Artificial Milk Formula or any source of DHA

Exclusion Criteria:

1. Age above 25 years.
2. Adult patients from 15 years to 25 years who feed on any Artificial Milk Formula or any source of DHA ..

Ages: 1 Day to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Newborn Infants and children feeding on Breast Milk or Artificial Milk Formula in the range from birth to about 15 years of age would be examined and followed between March 2020 and October 2021 and compare their rates of Covid-19 infection, hospitalization and complications with the rates of the Control Groups
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Susceptibility for COVID-19. | March2020 - October 2021
  Did infants and children who were fed breast milk or artificial milk formula have a lower risk of infection with Covid-19? in comparison with the control groups

SECONDARY OUTCOMES:
Severity for COVID-19. | March2020 - October 2021
  Did infants and children with COVID-19 who were fed breast milk or artificial milk formula have a lower chance of illness severity and requiring intensive care support or not in comparison with the control groups, ?
Mortality | March2020 - October 2021
  In comparison to the control groups, did newborns and children with COVID-19 who were fed breast milk or artificial milk formula have a reduced mortality rate?
Care and Critical Care | March2020 - October 2021
  Did infants and children with COVID-19 feeding on Breast Milk or Artificial Milk Formula have a shorter Length of hospitalization and stay in the ICU in comparison with the control groups
Resolution of fever | March2020 - October 2021
  In comparison to the control groups, did COVID-19-infected infants and children who were fed breast milk or artificial milk formula have a faster resolution of fever and did not require advanced fever management?
Percentage of children requiring intensive care support | March2020 - October 2021
Clinical symptoms of children | March2020 - October 2021

CONTACTS AND LOCATIONS:
Overall Officials: Dr Mahmoud R Elkazzaz, M.Sc of Biochemistry, Principal Investigator — Faculty of Science Damietta University; Dr Amr K Ahmed, Principal Investigator — Ministry of Health, Saudia Arabia

REFERENCES:
- See also: Natural phytochemicals, Phenformin, and Docosahexaenoic acid (DHA) as a Novel Inhibitors of IL-6 and ACE2 receptors, a Therapeutic Strategy for targeting COVID-19 Cell Entry and Cytokine Storm. An insilico Approach — https://www.researchsquare.com/article/rs-918251/v1